CLINICAL TRIAL: NCT06154811
Title: Predicting Extubation Outcomes in Mechanically Ventilated Patients Using PW-TDI Diaphragmatic Kinematics and Traditional Ventilation Parameters: A Prospective Study
Brief Title: Exploring the Use of Pulse Tissue Doppler in Predicting Extubation Success in Mechanically Ventilated Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Sponsor
Other Study IDs: 269089632
Record Dates: First submitted 2023-11-26; First posted 2023-12-04 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Airway Extubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Extubation Success Group: Extubation success is defined as the successful completion of a Spontaneous Breathing Trial (SBT) and the maintenance of spontaneous breathing without respiratory distress for at least 48 hours, without the need for non-invasive or invasive ventilation.
- Extubation Failure Group: Extubation failure is defined as successful Spontaneous Breathing Trial (SBT) but an inability to sustain independent breathing for more than 48 hours without non-invasive or invasive ventilation.

SUMMARY:
Determining the appropriate extubation timing for mechanically ventilated patients is a critical issue in the Intensive Care Unit (ICU). Early or delayed extubation may prolong mechanical ventilation and ICU stay, leading to an increased mortality rate. Currently, extubation timing relies solely on the Spontaneous Breathing Trial (SBT), but its reliability is relatively low, with a extubation failure rate ranging from 10% to 40%. Therefore, accurately predicting potential post-extubation issues and early identification of reasons for SBT trial failure are crucial for improving patient outcomes. Commonly used parameters for assessing readiness for extubation do not fully reflect organ dysfunction, and the investigators plan to utilize comprehensive techniques, including bedside lung and diaphragm ultrasound parameters, to enhance the accuracy of predicting extubation outcomes in patients who pass the SBT trial.

DETAILED DESCRIPTION:
All patients included in the study underwent a spontaneous breathing trial (SBT) using pressure support ventilation (PSV) strategy. This strategy employed pressure support(PS)≤9 cmH2O and positive end-expiratory pressure (PEEP)≤5 cmH2O. The duration of the trial was 30 minutes, and the FiO2 level was set at the same level (≤0.5) used during mechanical ventilation. After successful completion of the spontaneous breathing trial (SBT), ultrasound images were promptly acquired, and the Rapid Shallow Breathing Index (RSBI) was calculated based on the values displayed by the ventilator . Simultaneously, the Acute Physiology and Chronic Health Evaluation II (APACHE II) score was computed and recorded. The decision to extubate, made by the attending physician (unaware of the ultrasound examination parameters), was based on clinical judgment. The primary endpoint event was extubation failure, defined as successful completion of SBT but an inability to sustain spontaneous breathing for more than 48 hours without noninvasive or invasive ventilation support.

ELIGIBILITY:
Inclusion Criteria:

* Patients were enrolled if participants had been intubated and mechanically ventilated for more than 24 hours and were ready for participants first SBT according to ICU weaning criteria.

Exclusion Criteria:

* paralytic drugs taken within 24 hours prior to the trial;
* diagnosis of diaphragmatic paralysis or paradoxical movement of the hemidiaphragm detected by ultrasound or poor imaging quality;
* Pregnancy;
* Ascites;
* age<18years;
* Post-thoracotomy;
* Existence of pneumothorax;
* presence of large pleural effusion, subcutaneous emphysema, flail chest or right-sided rib fractures;
* presence of neuromuscular diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From September 01, 2022, to December 30, 2024, continuously enroll patients admitted to both ICU and EICU who, due to various pathophysiological reasons, require mechanical ventilation for more than 24 hours and have successfully passed a spontaneous breathing trial.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Successful Removal of Endotracheal Tube | The patient undergoes a spontaneous breathing trial, and measurements are taken 30 minutes after the removal of the endotracheal tube.
  Extubation success is defined as the successful completion of a Spontaneous Breathing Trial (SBT) and the maintenance of spontaneous breathing without respiratory distress for at least 48 hours, without the need for non-invasive or invasive ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Liu, Master, Study Director — Affiliated Hospital of Jiangnan University
Locations (1):
- Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Within 60 days of publication, we will share research data, including but not limited to the Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF), Clinical Study Report (CSR), and Analytic Code. The aforementioned research data will be uploaded in the form of case record sheets to https://github.com/.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: within 60 days of publication
Access Criteria: individual patient data(IPD) Sharing Standards
  Purpose:
  Data is solely for lawful, scientific research, not commercial or illegal use.
  Compliance:
  Usage complies with regulations, ethics, privacy principles.
  Research Proposal:
  Utilizing researchers submit detailed proposals.
  Ethical Review:
  Proposals need ethics committee approval.
  Data Security:
  Researchers ensure secure data handling.
  De-identification:
  Data provided is de-identified for privacy.
  Reporting Obligations:
  Researchers report progress and share results.
  Sharing Plan Updates:
  Data providers can update plans.
  Collaboration Opportunities:
  Data providers may collaborate on analysis, publications.
  Legal Responsibilities:
  Researchers follow legal regulations, preventing misuse.